CLINICAL TRIAL: NCT03638193
Title: Study of Autologous T-cells Redirected to Mesothelin With a Chimeric Antigen Receptor in Patients With Metastatic Pancreatic Cancer
Brief Title: Study of Autologous T-cells in Patients With Metastatic Pancreatic Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen BinDeBio Ltd. (Industry)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017NJYY-Meso
Record Dates: First submitted 2017-11-14; First posted 2018-08-20 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CART-meso cells (Experimental): A single dose of CART-meso T cells will be administered intravenously.The dose is 1-3×10^7/m^2 CART positive cells(chort 1)or 1-3×10^8/m^2 CART positive cells(chort 2).
  Interventions: Biological: CART-meso cells

INTERVENTIONS:
Biological: CART-meso cells — CART-meso is a 2nd CAR, with mesothelin as target protein, 4-1BB as co- stimulator. The infusion will be scheduled to occur 3 (±1) days after a single dose of 1.5 grams/m^2 of cyclophosphamide, which will be administered according to standard procedures, Thereby enhancing the efficacy of anti-tumor, reducing the potential of side effects.

SUMMARY:
This is a study in which pancreatic cancer patients receive a immunotherapy with CART-meso cells administered at 3 days after one dose of cyclophosphamide. CART-meso cells are patients' own T cells lentivirally transduced to express anti-mesothelin scFv fused to TCRζ and 4-1BB costimulatory domains.The lymphodepletion with cyclophosphamide may prolong the persistence of CART cells.

DETAILED DESCRIPTION:
This study is being conducted to assess the safety and efficacy of immunotherapy with CART-meso cells in dose escalation design. The trial will begin in Cohort 1 and progress to Cohorts 2, depending upon dose limiting toxicity (DLT) assessment .

Subjects will be enrolled serially, but infusions will be staggered to allow assessment of DLTs for determination of cohort progression, expansion, or dose de-escalation.

Cohort 1 subjects will receive a single dose of 1-3x10^7 /m^2 lentiviral transduced CART-meso cells after conditioning chemotherapeutic regimen.

Cohort 2 subjects will receive a single dose of 1-3x10^8 /m^2 lentiviral transduced CART-meso cells cells after conditioning chemotherapeutic regimen.

Dose limiting toxicity is defined as any adverse reactions at level 3 or above that may be associated with CART-meso within 4 weeks after infusion.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Unresectable or metastatic pancreatic cancer
* Persistent cancer after at least one prior standard of care chemotherapy for advanced stage disease
* 18 - 70 years of age
* ECOG performance status of 0 or 1
* Life expectancy greater than 3 months
* Satisfactory organ and bone marrow function
* Meets blood coagulation parameters
* Male and Female subjects of reproductive potential agree to use approved contraceptive methods

Exclusion Criteria:

* Participation in a therapeutic investigational study within 4 weeks prior to the screening visit
* Anticipated need for systemic chemotherapy within 2 weeks before apheresis and infusion
* Active invasive cancer other than pancreatic cancer
* HIV, HCV, or HBV infections
* Active autoimmune disease requiring immunosuppressive therapy within 4 weeks prior to screening visit, with exception of thyroid replacement
* Ongoing or active infection
* Planned concurrent treatment with systemic high dose corticosteroids
* Patients requiring supplemental oxygen therapy
* Prior therapy with gene modified cells
* Previous experimental therapy with SS1 moiety, murine or chimeric antibodies
* History of allergy to murine proteins
* History of allergy or hypersensitivity to study product excipients (human serum albumin, DMSO, and Dextran 40)
* Clinically significant pericardial effusion, CHF, or cardiovascular condition that would preclude assessment of mesothelin induced pericarditis or that may worsen as a result of toxicities expected for this study
* Pregnant or breastfeeding women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-07-11 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Safety of CART-meso infusion: number of adverse events | 60 months
  Number of Adverse Events evaluated with NCI CTC AE, version 4.0[Safety evaluation]

SECONDARY OUTCOMES:
Clinical response of CART-meso | 60 months
  Number of patients with tumor response including overal remission ,complete ression,progression-free survival，progressive disease ,etc.
CAR-T cell detection | 60 months
  Detection of transferred T cells in peripheral blood or bone marrow using multi-parameter flow cytometer.

CONTACTS AND LOCATIONS:
Overall Officials: Jinfei CHEN, MD, PhD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China